CLINICAL TRIAL: NCT05552183
Title: A Phase 1, Open-label, Multiple-dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Pacritinib in Subjects With Varying Degrees of Hepatic Impairment Compared to Healthy Subjects
Brief Title: Study to Evaluate the Safety, Tolerability, and PK of Pacritinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAC110
Record Dates: First submitted 2022-09-13; First posted 2022-09-23 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Hepatic Impairment
Keywords: Pacritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Moderate Hepatic Impairment (Experimental): Subjects with moderate hepatic impairment based on Child-Pugh Class B score of 7-9 will receive 14 days of 200 mg BID pacritinib.
  Interventions: Drug: oral dose of 200 mg pacritinib twice daily (BID)
- Severe Hepatic Impairment (Experimental): Subjects with severe hepatic impairment based on Child-Pugh Class C score of 10-15 will receive 14 days of 200 mg BID pacritinib.
  Interventions: Drug: oral dose of 200 mg pacritinib twice daily (BID)
- Normal Hepatic Function (Experimental): Healthy subjects who have normal hepatic function with age (± 10 years; ≥ 18 years old and ≤ 85 years old), BMI (±20%), and sex, matching with the moderate and severe hepatic impairment cohorts will receive 14 days of 200 mg BID pacritinib.
  Interventions: Drug: oral dose of 200 mg pacritinib twice daily (BID)

INTERVENTIONS:
Drug: oral dose of 200 mg pacritinib twice daily (BID) — Subjects will receive 200 mg BID pacritinib for 14 days.

SUMMARY:
This is a Phase 1 study designed to assess the effect of hepatic insufficiency on the PK of pacritinib by study of 14-day BID dosing of pacritinib in subjects with moderate and severe hepatic impairment compared to healthy matched control subjects with normal liver function. Safety and tolerability of multiple day dosing of pacritinib in the subject populations will also be evaluated.

DETAILED DESCRIPTION:
This is a Phase 1, multi-center, open-label, multiple-dose, parallel-group study designed to assess the effect of hepatic insufficiency on the PK of 200 mg BID pacritinib. A total of approximately 22 to 32 subjects are planned, with approximately 8 moderate hepatically impaired subjects, approximately 6 to 8 severe hepatically impaired subjects, and approximately 8 to 16 healthy subjects with normal hepatic function. The primary objective of this study is to characterize and compare the steady-state PK profile of multiple doses (14 days) of 200 mg BID pacritinib in the study population, and the secondary objective is to evaluate the safety and tolerability of multiple doses (14 days) of 200 mg BID pacritinib. The study will consist of a screening period (Day -28 to Day -2), check-in (Day -1), a confinement period including treatment period (Day 1 through Day 14) and post-treatment period (Day 15 through Day 20), followed by a discharge visit (Day 21), and an EOS follow-up telephone call (Day 44). Serial blood samples for PK analysis of pacritinib will be collected pre dose through Day 21 at protocol-specified timepoints CK 18 will be collected . Safety and tolerability will be assessed by AEs, clinical laboratory tests, vital will occur 4 and 24 hours after the AM dose on Day 1, Day 10, Day 12, and Day 14 signs, ECGs, and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent.
2. Able to communicate well with the investigator and understands and agrees to comply with all protocol requirements.
3. Is male or female ≥18 to ≤85 years of age, inclusive, at screening.
4. Has a BMI 18.0 to 42.0 kg/m2, inclusive, at screening.
5. Female subjects of childbearing potential must be surgically sterile, or postmenopausal, or agree use an acceptable method of birth control from the time of ICF or 10 days prior to check-in and until 30 days after Day 21. Female subjects of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at check-in.
6. Male subjects with female partners of childbearing potential must be vasectomized, be willing to use an acceptable method of birth control, or to practice abstinence during the study from check-in until 90 days following Day 21.
7. Male subjects must refrain from sperm donation from check-in until 90 days following Day 21.

   Additional Inclusion Criteria for Subjects with Hepatic Impairment Only:
8. Has chronic (>6 months) and stable hepatic impairment (ie, no acute episodes of illness within 30 days prior to screening due to deterioration of hepatic function) as assessed by a Child-Pugh classification score of moderate (7 to 9 points) or severe (10 to 15 points).
9. Is judged by the investigator to be in good general health, as determined by medical history, clinical laboratory assessments, vital sign measurements, 12 lead ECG results, and physical examination findings, except for findings that, as judged by the investigator, are consistent with the subject's hepatic impairment or other stable concomitant medical conditions at screening and check-in.

   Additional Inclusion Criteria for Healthy Subjects Only:
10. Has normal hepatic function.
11. Must match a subject in Group 1 and/or Group 2, with respect to sex, age (±10 years), and BMI (±20%).
12. Is judged by the investigator to be in good general health, as determined by medical history, clinical laboratory assessments, vital sign measurements, 12 lead ECG results, and physical examination findings at screening and check-in.

Exclusion Criteria:

1. Has a history or clinical manifestations of a significant neurological, renal, cardiovascular, gastrointestinal, pulmonary, hematologic, immunologic, or psychiatric disease that would preclude study participation, as judged by the investigator.
2. Has any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs or which may jeopardize the subjects participation in the study. The investigator should be guided by evidence of any of the following:

   * History of inflammatory bowel disease
   * History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection (esophageal varix surgery is allowable)
   * Clinical evidence of pancreatic injury or pancreatitis
   * Evidence of urinary obstruction or difficulty in voiding at screening
3. Has a baseline seated systolic blood pressure >160 mm Hg or ≤90 mm Hg and a diastolic blood pressure of >100 mm Hg or ≤50 mm Hg, inclusive, at screening and check in unless deemed not clinically significant by the investigator, as approved by the sponsor.
4. Has a baseline seated pulse rate of <50 bpm or >100 bpm and/or an oral body temperature <35.0°C or >37.5°C when vital signs are measured at screening and check in.
5. Has a significant QT interval prolongation (QTcF of >480 msec) or other risks for QT prolongation at screening or check-in.
6. Has a history of being immunocompromised or has a positive serum test result for HIV types 1 or 2 antibodies at screening.
7. Has had a significant illness within the 2 weeks prior to check-in.
8. Has a history of alcoholism, drug abuse, or alcohol withdrawal within 3 months before screening, or excessive alcohol consumption (regular alcohol intake >21 units per week for male subjects and >14 units of alcohol per week for female subjects) (1 unit is equal to approximately ½ pint [200 mL] of beer, 1 small glass [100 mL] of wine, or 1 measure [25 mL] of spirits).
9. Is unable or unwilling to abstain from alcohol from 72 hours prior to check-in until Day 21.
10. Is unable or unwilling to abstain from caffeine, xanthine-containing beverages or food (eg, coffee, tea, chocolate, and caffeinated sodas, colas) from check in until Day 21.
11. Has consumed grapefruit, grapefruit juice, Seville oranges, or products containing any of these, from 7 days prior to check-in to the study site until Day 21.
12. Smokes >10 cigarettes daily and is unwilling to reduce to ≤5 daily from the time of screening through Day 21.
13. Is involved in strenuous activity or contact sports within 24 hours prior to check-in or during the study.
14. Has donated blood or blood products >450 mL within 30 days prior to the first dose of study drug.
15. Has used over-the-counter medications (except as prescribed by a physician or paracetamol [up to 2 g per day]), vitamins, or phyto-therapeutic/herbal/plant-derived preparations within 14 days of check-in.
16. Has used a potent CYP3A4 inducer within 30 days prior to check-in or used a potent CYP3A4 inhibitor within 15 days prior to check-in.
17. Has received treatment in another clinical study of an investigational drug (or medical device) or investigational vaccine within 30 days or 5 half-lives (whichever is longer) prior to check-in.
18. The subject has previously received pacritinib.
19. Has a known hypersensitivity to study drug (ie, allergy to pacritinib or any excipients or drugs similar to pacritinib).
20. Has had a recent bleeding event of Grade ≥2 within 3 months prior to first dose of study drug.
21. Has used antiplatelet or anticoagulant therapy within 14 days prior to check in with the exception of aspirin at doses ≤100 mg daily.
22. Has a history of heart failure with a New York Heart Association Class II or above.
23. Has a recent cardiac event of Grade ≥3 within 6 months prior to check in.
24. In the opinion of the investigator, the subject is not suitable for entry into the study.

    Additional Exclusion Criteria for Subjects with Hepatic Impairment Only:
25. Has fluctuating or rapidly deteriorating hepatic function, as indicated by recent history or worsening of clinical (ie, abdominal pain, nausea, vomiting, anorexia, or fever) and/or laboratory signs of hepatic impairment, as judged by the investigator.
26. Has symptoms or history of Stage II or worse degree of encephalopathy that would prohibit informed consent within 6 months before check-in, as judged by the investigator.
27. Has clinical evidence of ascites that requires paracentesis more frequently than every 3 weeks at screening or check-in.
28. Has a history of a surgical portosystemic shunt.
29. Has evidence of hepatorenal syndrome.
30. Has any of the following laboratory results:

    * Estimated serum creatinine clearance (Cockcroft-Gault) <50 mL/min
    * Absolute neutrophil count <1500 cells/mm3
    * Platelet count <30,000 cells/mm3
    * Hemoglobin <9 g/dL
    * Activated partial thromboplastin time, international normalized ratio, partial thromboplastin time, or prothrombin time clinically significant per investigator discretion.
31. Has evidence of progressive liver disease (as available within the last 4 weeks, including the time period between screening and check-in) as indicated by liver transaminases, alkaline phosphatase, and gamma-glutamyl transpeptidase, as judged by the investigator.
32. Has evidence of active acute or chronic hepatitis B virus.
33. Has a positive test result for drugs of abuse (except for positive results associated with prescription medications that have been reviewed and approved by the investigator) or positive alcohol urine or breath test at screening or check-in. A positive tetrahydrocannabinol result at screening will not be exclusionary, but must be negative at check-in.
34. Has a urinalysis with any result outside the normal range and deemed clinically significant by the investigator. Results deemed not clinically significant by the investigator in consultation with the sponsor may be allowed.
35. Has initiated any otherwise allowable prescription or over-the-counter medications within 15 days of check-in. Some of these medications may have to be discontinued 12 to 48 hours before study drug dosing, or earlier. As medication regimens vary and cannot be predicted, each subject will be discussed with the sponsor individually. The dose of an approved medication must remain stable from 7 days before study drug dosing and throughout the study.

    Additional Exclusion Criteria for Healthy Subjects Only:
36. Has a positive test result for hepatitis B surface antigen and/or hepatitis C virus antibodies.
37. Any screening or check-in laboratory results outside the normal range and deemed clinically significant. Results outside the normal range and deemed not clinically significant by investigator, in consultation with the sponsor, are allowable.
38. Has used any prescription medication within 30 days prior to check in.
39. Activated partial thromboplastin time, international normalized ratio, partial thromboplastin time, or prothrombin time > 1.5 × ULN.
40. Has a positive test result for drugs of abuse or positive alcohol urine or breath test prior to the first dose of study drug.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
PK | Day 1- (Day 1: Cmax)
  To characterize and compare the steady-state PK profile of multiple doses (14 days) of 200 mg BID pacritinib in subjects with moderate and severe hepatic impairment with that of healthy matched control subjects with normal liver function.
PK | Day 1(Day 1: Tmax)
  To characterize and compare the steady-state PK profile of multiple doses (14 days) of 200 mg BID pacritinib in subjects with moderate and severe hepatic impairment with that of healthy matched control subjects with normal liver function.
PK | Day 1( AUC0-12)
  To characterize and compare the steady-state PK profile of multiple doses (14 days) of 200 mg BID pacritinib in subjects with moderate and severe hepatic impairment with that of healthy matched control subjects with normal liver function.
PK | Day 14: Cmax,
  To characterize and compare the steady-state PK profile of multiple doses (14 days) of 200 mg BID pacritinib in subjects with moderate and severe hepatic impairment with that of healthy matched control subjects with normal liver function.
PK | Day 14: Tmax,
  To characterize and compare the steady-state PK profile of multiple doses (14 days) of 200 mg BID pacritinib in subjects with moderate and severe hepatic impairment with that of healthy matched control subjects with normal liver function.
PK | Day 14 t1/2
  To characterize and compare the steady-state PK profile of multiple doses (14 days) of 200 mg BID pacritinib in subjects with moderate and severe hepatic impairment with that of healthy matched control subjects with normal liver function.
PK | Day 14 CL/F
  To characterize and compare the steady-state PK profile of multiple doses (14 days) of 200 mg BID pacritinib in subjects with moderate and severe hepatic impairment with that of healthy matched control subjects with normal liver function.
PK | Day 14 AUC0 t
  To characterize and compare the steady-state PK profile of multiple doses (14 days) of 200 mg BID pacritinib in subjects with moderate and severe hepatic impairment with that of healthy matched control subjects with normal liver function.
PK | Day 14 AUC0 -12
  To characterize and compare the steady-state PK profile of multiple doses (14 days) of 200 mg BID pacritinib in subjects with moderate and severe hepatic impairment with that of healthy matched control subjects with normal liver function.
PK | Day 14 λZ,
  To characterize and compare the steady-state PK profile of multiple doses (14 days) of 200 mg BID pacritinib in subjects with moderate and severe hepatic impairment with that of healthy matched control subjects with normal liver function.
PK | Day 14 Vz/F
  To characterize and compare the steady-state PK profile of multiple doses (14 days) of 200 mg BID pacritinib in subjects with moderate and severe hepatic impairment with that of healthy matched control subjects with normal liver function.
PK | Day 14 f/u
  To characterize and compare the steady-state PK profile of multiple doses (14 days) of 200 mg BID pacritinib in subjects with moderate and severe hepatic impairment with that of healthy matched control subjects with normal liver function.
PK | Day 14 ARCmax
  To characterize and compare the steady-state PK profile of multiple doses (14 days) of 200 mg BID pacritinib in subjects with moderate and severe hepatic impairment with that of healthy matched control subjects with normal liver function.
PK | Day 14 ARAUC0-12
  To characterize and compare the steady-state PK profile of multiple doses (14 days) of 200 mg BID pacritinib in subjects with moderate and severe hepatic impairment with that of healthy matched control subjects with normal liver function.

SECONDARY OUTCOMES:
Incidence of adverse events | Day 1-44
  Safety and tolerability of pacritinib, including monitoring of adverse events (AEs); an AE is any untoward medical occurrence in a study subject administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage
Incidence of clinical laboratory abnormalities | Day 1-21
  Safety and tolerability of pacritinib, including hematology, coagulation, chemistry, and urinalysis parameters
Incidence of vital sign abnormalities | Day 1-21
  Safety and tolerability of pacritinib, including monitoring of blood pressure, heart rate, respiratory rate, and body temperature
Incidence of ECG abnormalities | Day1-21
  Safety and tolerability of pacritinib, including monitoring of RR interval, PR interval, QRS width, QT interval, and QTcF
Incidence of physical examination abnormalities | Day 1-21
  Safety and tolerability of pacritinib, including monitoring for abnormalities on physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Buckley, Study Director — Sobi, Inc.
Locations (2):
- United States (2):
  - Site 2, Orlando, Florida
  - Site 1, San Antonio, Texas